CLINICAL TRIAL: NCT05647577
Title: Prevalence and Risk Factors Associated With Cardiac Comorbidity in Inflammatory Arthritis - A Prospective Cohort Study
Brief Title: The Relationship Between Inflammatory ARTritis and CArdiac DIseAse
Acronym: ARTCADIA
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Tor Biering-Sørensen, Professor in Translational Cardiology and Pragmatic Randomized Trials, University Hospital, Gentofte, Copenhagen
Other Study IDs: H-20023771
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Inflammatory Arthritis; Rheumatoid Arthritis; Spondylitis, Ankylosing; Axial Spondyloarthritis; Spondyloarthritis; Heart Failure; Ischemic Heart Disease; Valvular Heart Disease; Left Ventricular Systolic Dysfunction; Heart Failure, Systolic; Heart Failure, Diastolic; Myocardial Infarction; Myocardial Dysfunction; Cardiac Disease; Stroke
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Axial Spondyloarthritis; Spondylarthritis; Heart Failure; Myocardial Ischemia; Heart Valve Diseases; Ventricular Dysfunction, Left; Heart Failure, Systolic; Heart Failure, Diastolic; Myocardial Infarction; Heart Diseases; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — whole blood and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inflammatory arthritis patients: Patients with an confirmed diagnosis of rheumatoid arthritis or axial spondyloarthritis.
- Participants from the general population: Patients with inflammatory arthritis will be compared to community-dwelling individuals from the 4th and 5th examination round from the Copenhagen City Heart Study (ClinicalTrials.gov identifier NCT02993172, I-Suite no. 03741, National Committee on Health Research Ethics approval HEH-2015-045).

SUMMARY:
The goal of this prospective cohort study is to investigate cardiac comorbidity in a random sample of approximately 1200 patients from a population of outpatients with rheumatoid arthritis and axial spondyloarthritis referred to collectively as inflammatory arthritis (IA). The main questions it aims to answer are:

* Using conventional echocardiography, the investigators aim to determine the prevalence of overt and asymptomatic cardiac dysfunction in a large random sample of outpatients with IA. Cardiac dysfunction will be evaluated by echocardiography and cardiac biomarkers (NT-pro-BNP, hs-TNT and hs-CRP).
* In patients without known heart disease: Using 2, 5 and 10 year follow-up, the investigators aim to examine if advanced echocardiography can be used to detect early signs of heart disease by investigating the clinical significance of adding deformation measures - alone and in combination with selected biomarkers - to conventional risk factors in the cardiac risk assessment of patients with IA

Participants will undergo an echocardiographic examination in combination with a general health assessment including obtainment of cardiac biomarkers and a electrocardiogram.

Using advanced echocardiography - Tissue Doppler Imaging, 2- dimensional speckle tracking echocardiography, 3D-echocardiography and 3-dimensional speckle tracking echocardiography - the investigators also aim to compare myocardial deformation parameters of patients with IA to a gender and age matched control group without IA from the Copenhagen City Heart Study.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a diagnosis of with a confirmed diagnosis of rheumatoid Arthritis or axial spondyloarthritis

Exclusion Criteria:

* Persons not able to cooperate
* Persons unable understand and sign "informed consent"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to approximate a random sample as accurate as possible, all patients with a diagnosis of rheumatoid Arthritis or axial spondyloarthritis followed in DANBIO in the capital region of Denmark will be eligible to participate. DANBIO is a nationwide registry of patients with rheumatoid Arthritis or axial spondyloarthritis and is approved as a clinical quality registry by the Danish National Board of Health in 2006.
Sampling Method: Probability Sample
Enrollment: 1285 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2033-03-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality | 2-year follow-up
Cardiovascular mortality | 5-year follow-up
Cardiovascular mortality | 10 year outcome
Admission with congestive heart failure | 2-year follow-up
Admission with congestive heart failure | 5-year follow-up
Admission with congestive heart failure | 10 years
Myocardial infarction | 2-year follow-up
Myocardial infarction | 5-year follow-up
Myocardial infarction | 10 years
Revascularization | 2-year follow-up
  Percutaneous coronary intervention or coronary artery bypass graft
Revascularization | 5-year follow-up
  Percutaneous coronary intervention or coronary artery bypass graft
Revascularization | 10-year follow-up
  Percutaneous coronary intervention or coronary artery bypass graft
Incident Heart Failure | 2-year follow-up
Incident Heart Failure | 5-year follow-up
Incident Heart Failure | 10-year follow-up
Incident valvular disease | 2-year follow-up
Incident valvular disease | 5-year follow-up
Incident valvular disease | 10-year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology | Center for Translational Cardiology and Pragmatic Randomized Trials (CTCPR) Cardiovascular Non-Invasive Imaging Research Laboratory (CIRL), Hellerup, Denmark